CLINICAL TRIAL: NCT03128372
Title: Validation of Next Generation INVOS NIRS Cerebral and Tissue Oximeter to Measure Cerebral and Somatic Tissue Oxygen Saturation in Healthy Volunteers
Brief Title: Validation of Next Generation Cerebral and Tissue Oximeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MDT16010MAVJB3
Record Dates: First submitted 2017-04-05; First posted 2017-04-25 (Actual); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Desaturation (Experimental): Volunteers undergo oxygen desaturation in order to determine the accuracy of the device over a clinical range of oxygen saturations 70 - 100%.
  Interventions: Device: Desaturation

INTERVENTIONS:
Device: Desaturation — The delivered gas mixture will be adjusted to decrease the displayed saturation of peripheral oxygen. Each desaturation steps are of approximately 5 minutes duration with reduction in pulse oximeter oxygen saturation from 100 to 70%.
  Other Names: Cerebral and Tissue Oximeter

SUMMARY:
This is a validation study of a near-infrared spectroscopy (NIRS) device designed to measure the cerebral tissue oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects between the ages of 18 to ≤46 years;
2. Completion of a health screening for a medical history by a licensed physician, nurse practitioner or physician assistant;
3. Minimum weight 40kg;
4. BMI within range 18.0 - 30.0.

Exclusion Criteria:

1. Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain) [self-reported];
2. Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported];
3. Taking any medication other than birth control [self-reported];
4. Is currently participating in, or has recently participated in (discontinued within 30 days prior to the hypoxia procedure for this study) in an investigational drug, device, or biologic study [self-reported];
5. Has a negative Allen's Test to confirm non-patency of the collateral artery [clinical assessment by PI or delegate];
6. Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported];
7. Is female with a positive pregnancy test [serum or urine], or is female and is unwilling to use effective birth control between the time of screening and study procedure or is breastfeeding;
8. Has anemia [lab values specific for gender];
9. Has a history of sickle cell trait or thalassemia [self-reported];
10. Has an abnormal hemoglobin electrophoresis test [lab measurement];
11. Has a positive urine cotinine test or urine drug screen or oral ethanol test [POC testing];
12. Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate];
13. Has a clinically significant abnormal ECG [assessment by PI or delegate];
14. Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
15. Has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co-oximetry]

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Katilius, Study Director — Medtronic
Locations (1):
- Duke University Hospital, HPPL, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desaturation
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Desaturation
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 19
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Validated the Next Generation Oximeter
Description: Cerebral overall mean bias (percentage saturation) defined as the average of the differences between the regional saturation (rSO2) value and (fSO2) value obtained from simultaneous arterial and jugular venous blood samples. Cerebral trending is defined as the measurement of changes in regional saturation (rSO2) under conditions of changing fSO2. Cerebral trending mean bias is the average difference between changes in rSO2 values compared against changes in fSO2. Somatic trending mean bias is defined the same as Cerebral trending mean bias except for the location of measurement on the subjects and for Somatic trending mean bias, rS02 was compared to rSO2 on a commercially-available regional oximetry monitor. The smaller value the better performance.
Time Frame: Data collected from individual participant over 4 hour timeframe.
Measure: Mean (Standard Deviation); unit: Percentage saturation
Arm/Group | Desaturation
Number analyzed (Participants) | 32
Percentage saturation
  Cerebral Overall Mean Bias | 1.22 (5.92)
  Cerebral Overall Trending Mean Bias | 0.83 (3.08)
  Somatic Overall Trending Mean Bias | 0.09 (1.73)

ADVERSE EVENTS:
Time Frame: 48 hours post study procedure (desaturation)
Arm/Group | Desaturation
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desaturation (N=32)
Vasovagal episode (Nervous system disorders) | 1 (1)
Clavicular pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03128372/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT03128372/SAP_001.pdf